CLINICAL TRIAL: NCT06305442
Title: Efficacy of Microbiota-Directed Food in Children With Moderate Acute Malnutrition in Dhaka, Bangladesh
Brief Title: Microbiota Directed Food for Children With Moderate Acute Malnutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-24031
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-02

CONDITIONS: Moderate Acute Malnutrition
Keywords: Microbiota Directed Food; Gut microbiota; MAM; Bangladesh
MeSH Terms: interventions — milk-derived factor

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel group, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiota Directed Food (MDF) (Experimental): Each participant will receive 12 weeks of MDF supplement. After finishing the intervention phase, he/she will be followed-up for a 12-week period.
  Interventions: Dietary Supplement: Microbiota-Directed Food
- Ready-to-Use Supplementary Food (RUSF) (Active Comparator): Each participant will receive 12 weeks of RUSF supplement. After finishing the intervention phase, he/she will be followed-up for a 12-week period.
  Interventions: Dietary Supplement: Ready-to-Use Supplementary Food

INTERVENTIONS:
Dietary Supplement: Microbiota-Directed Food — MDF is a microbiota directed food for malnourished children aged 6 months and above. It is in sachet form. The sachet contains 92 gm of supplements and provides approximately 506 kcal.
  Other Names: MDF
  Arms: Microbiota Directed Food (MDF)
Dietary Supplement: Ready-to-Use Supplementary Food — RUSF is standard ready-to-use supplementary food for MAM children aged 6 months and above.
  Other Names: RUSF
  Arms: Ready-to-Use Supplementary Food (RUSF)

SUMMARY:
Moderate acute malnutrition (MAM) refers to a condition characterized by a significant deficit in weight-for-length measurements in children aged 6 to 59 months. It is a crucial public health concern with detrimental effects on child growth, development, and overall well-being. Addressing MAM is crucial to prevent its progression to severe acute malnutrition (SAM) and to ensure healthy child development. To meet the nutritional requirement of MAM children, icddr,b have come up with a novel intervention named microbiota-directed food (MDF), a ready-to-use supplementary food. The investigator propose this efficacy trial to establish the evidence on the effect of this novel intervention on ponderal growth, microbial and proteomic recovery among the children with MAM in comparison to the standard RUSF.

DETAILED DESCRIPTION:
Burden: Moderate acute malnutrition (MAM) refers to a condition characterized by a significant deficit in weight-for-length measurements in children aged 6 to 59 months. It is a crucial public health concern with detrimental effects on child growth, development, and overall well-being. Addressing MAM is crucial to prevent its progression to severe acute malnutrition (SAM) and to ensure healthy child development. MAM affects a significant number of children globally, particularly in low- and middle-income countries where malnutrition is prevalent. According to the 2022 Bangladesh Demographic and Health Survey (2022 BDHS), 24% of children under the age of 5 are stunted, while 11% are wasted. The prevalence of worldwide MAM children is higher than that of children with SAM and 31.3 million under 5 children (~70%) was moderately wasted among all those children who were acutely malnourished in 2022. MAM children are found to be suffering from relative gut microbial immaturity, which is related to their growth faltering. Ready-to-use supplementary food (RUSF) is a key component of the outpatient treatment of MAM in community-based management. RUSF, being a ready-to-use food, does not require preparation or refrigeration and provides the necessary nutrients and energy for recovery from MAM.

Knowledge gap: Researchers at icddr,b in collaboration with Washington University in St. Louis, have developed a Microbiota-Directed Complementary Food (MDCF) formulation (based on locally available food ingredients) that has the potential to repair the gut microbiota of children with malnutrition. Results from a recently conducted study of MDCF on Bangladeshi children suffering from MAM showed that the children who received the food exhibited significantly faster rates of ponderal growth compared to those treated with a standard ready-to-use supplementary food (PR#18073). Early evidence, however, is limited to a small sample of children with MAM.

Relevance: To meet the nutritional requirement of MAM children, icddr,b have come up with a novel intervention named microbiota-directed food (MDF), a ready-to-use supplementary food by modifying the original MDCF recipe to meet the nutritional requirement of MAM children as well as to make it align with the existing WHO/UNICEF specifications for a nutritional intervention for treating acute malnutrition. The proposed formulation of MDF with adequate calorie content will improve the nutritional status by modulating and improving the gut microbial dysbiosis that is present in MAM children. Therefore, the investigator propose this efficacy trial to establish the evidence on the effect of this novel intervention on ponderal growth, microbial and proteomic recovery among the children with MAM in comparison to the standard RUSF.

Hypothesis (if any):

The locally developed MDF would be proven beneficial in nutritional recovery, repairing microbiota and restoring plasma biomarkers of healthy growth when compared to standard RUSF among children suffering from MAM.

Objectives:

Primary objectives:

•To assess the efficacy of MDF in improving the weight-for-length Z score (WLZ) of MAM children

Secondary:

* To investigate the efficacy of MDF in repairing the microbiota of MAM children
* To measure the efficacy of MDF in improving the Weight-for-Age Z-score (WAZ) in children with MAM
* To measure the efficacy of MDF in improving the Length-for-Age Z-score (LAZ) in children with MAM
* To explore and validate the impact of MDF supplement in restoring plasma and fecal biomarkers
* To monitor the change produced by MDF in rebalancing the body composition (fat mass % and fat-free mass %)
* To explore the efficacy of MDF in improving the cognitive, motor, and language function of MAM children

Methods:

Study Design: This study will be a double-blind, randomized controlled trial.

Participants: The trial will recruit 6-24-months-old children with Moderate Acute Malnutrition

Study Site: Bauniabadh and the adjacent slum area of Mirpur in Dhaka city.

Sample Size: 230; 2 arms; 115 per arm)

Intervention: Children in one arm will receive the MDF, and the children in the control arm will receive the conventional RUSF.

The children will receive intervention for 12 weeks with either the MDF or RUSF.

* 6-24-months children with MAM - 12 weeks intervention with MDF + 12 weeks follow up
* 6-24-months children with MAM - 12 weeks intervention with RUSF + 12 weeks follow up

Study Procedure Screening, and enrolment of study participants will be done in Bauniabadh and the adjacent slum area of Mirpur in Dhaka city. Initially 6-24-months-old children will be screened by the study health workers. Parents of eligible children who meet the inclusion criterion will be approached about enrolment into the study. A trained Field Research Assistant will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enroll the child in the study. After acquiring consent from the parents, at the beginning of the study, information will be sought on the demographic characteristics (families' wealth, standard of housing, family structure, home environment, parental characteristics etc.). Morbidity data will be collected weekly during the intervention period, and biweekly in the follow-up phase.

In this study, nutritional status will be assessed through anthropometry, comparing with WHO growth reference standards. BIA is a method of assessing body composition by measuring body fat in relation to lean body mass. It is an integral part of a health and nutrition assessment. BIA will be used to measure total fat and fat-free mass before and after treatment. This non-invasive test simply involves the placement of electrodes on the person's hand and foot. A low-level, imperceptible electrical current is sent through the body. The flow of the current is affected by the amount of water in the body. The device measures how this signal is impeded through different types of tissue as it passes through the body and provides estimates of body water from which body fat is calculated.

A food frequency questionnaire will be used to collect data on Infant and Young Child Feeding (IYCF) practices. Food frequency data will be evaluated using the Minimum Acceptable Diet indicator as it meets standards for both minimum dietary diversity and minimum meal frequency.

The Bayley Scales of Infant and Toddler Development (BSID-IV) will be used to assess the early childhood development (cognitive, motor, and language development) before and after the intervention. The Caregiver Reported Early Development Instruments (CREDI) long form, developed by Harvard University, will also be used in this study (21).

Blood samples will be collected before, after the intervention/treatment, and at the end of the follow-up period for measuring haemoglobin, serum protein (total protein and albumin), thiamine, zinc, vitamin B12, vitamin D, and folate levels.

Non-diarrheal stool samples will be collected at enrolment, then monthly during the intervention and follow-up phase from all the participants for measuring biomarkers of gut inflammation and assessment of the composition of gut microbiota and features of the microbiome.

Oral swab samples will be collected by using commercial kit from each child at enrolment, after the intervention/treatment, and at the end of the follow-up period for measuring microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s) willing to sign consent form
2. Children aged 6-24 months
3. WLZ score <-2 to ≥-3 and/or MUAC ≥115 mm to <125 mm without bilateral pedal edema at the time of randomization

Exclusion Criteria:

1. Medical conditions: Malnourished children with complications requiring acute phase treatment in a hospital, children with tuberculosis or any chronic illness(es).
2. Any congenital/acquired disorder affecting growth, i.e., known case of trisomy-21 or cerebral palsy; children on an exclusion diet for the treatment of persistent diarrhea; having known history of soy, peanut or milk protein allergy
3. Severe anaemia (< 8 gm/dl)
4. Antibiotic use (within last 7 days before the onset of intervention)
5. Receiving concurrent treatment for another condition
6. children participating in other food intervention program

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change in Weight-for-Length Z-score (WLZ) | Baseline to 12 weeks of intervention followed by 12 weeks of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement before enrolment, then biweekly till completion of intervention and monthly during 12 weeks follow up.

SECONDARY OUTCOMES:
Microbial community repair | Baseline to 12 weeks of intervention followed by 12 weeks of follow-up
  Non-diarrheal stool samples will be collected at enrolment, then monthly during the intervention and follow-up phase from all the participants for assessment of the composition of gut microbiota and features of the microbiome.
  Oral swab samples will be collected by using commercial kit from each child at enrolment, after the intervention/treatment, and at the end of the follow-up period for measuring microbiota.
Validated plasma and faecal biomarkers of health status (prioritized Luminex/ELISA panel including mediators of growth, systemic inflammation, gut inflammation/entero-pathogen burden) | Baseline to 12 weeks of intervention followed by 12 weeks of follow-up
  Blood samples will be collected before, after the intervention/treatment, and at the end of the follow-up period.
  Non-diarrheal stool samples will be collected at enrolment, then monthly during the intervention and follow-up phase from all the participants for measuring biomarkers of gut inflammation.
Mean change in Weight-for-Age Z-score (WAZ) | Baseline to 12 weeks of intervention followed by 12 weeks of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement before enrolment, then biweekly till completion of intervention and monthly during 12 weeks follow up.
Mean change in Length-for-Age Z-score (LAZ) | Baseline to 12 weeks of intervention followed by 12 weeks of follow-up
  In this study, nutritional status will be assessed through anthropometric measurement before enrolment, then biweekly till completion of intervention and monthly during 12 weeks follow up.
Mean change in body composition (% body fat mass and % fat-free mass) | Baseline to 12 weeks of intervention
  In this study, nutritional status will be also assessed through Bioelectrical impedance at enrolment and after completion of intervention
Bayley Scales of early childhood development (cognitive, motor, language development) | Baseline to 12 weeks of intervention
  The Bayley Scales of Infant and Toddler Development (BSID-IV) will be used to assess the early childhood development (cognitive, motor, and language development) before and after the intervention. The Bayley-4 utilizes standard scores to assess a child's developmental progress compared to their age peers. Derived from individual raw scores, standard scores (with a mean of 100 and standard deviation of 15) offer a standardized metric for comparisons across Bayley-4 domains. The interpretation of standard scores on the Bayley-4 involves comparing an individual child's scores to the normative data provided in the test manual. Scores falling within one standard deviation (85-115) are considered within the average range, while scores below 85 in any domain may indicate potential developmental delays or concerns in that respective domain. Conversely, scores above 115 may suggest advanced development in that respective domain. Higher scores will mean better development.

CONTACTS AND LOCATIONS:
Overall Officials: Ishita Mostafa, BDS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Mirpur Study site, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No